CLINICAL TRIAL: NCT00293020
Title: An Open Label, Long-term Treatment Evaluation of the Safety of BEMA™ Fentanyl Use for Breakthrough Pain in Cancer Subjects on Chronic Opioid Therapy
Brief Title: Study of the Safety of BEMA™ Fentanyl Use for Breakthrough Pain in Cancer Subjects on Chronic Opioid Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEN-202
Record Dates: First submitted 2006-02-15; First posted 2006-02-17 (Estimated); Results first posted 2012-10-05 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-09

CONDITIONS: Pain; Cancer
Keywords: Breakthrough Pain in Cancer Patients
MeSH Terms: conditions — Pain; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): BEMA Fentanyl
  Interventions: Drug: BEMA Fentanyl

INTERVENTIONS:
Drug: BEMA Fentanyl — buccal soluble film; 200, 400, 600, 800, 1200 mcg fentanyl; up to 4 times daily
  Other Names: bioerodible mucoadhesive system

SUMMARY:
The purpose of this study is to evaluate the safety of BEMA fentanyl at any dose in the management of breakthrough pain in cancer subjects on background opioid therapy. The standard of care for these breakthrough pain episodes is a rapid onset, short acting analgesic with minimal associated sleepiness. Oral morphine, oxycodone and hydromorphone are routinely used, but because of slow and variable oral absorption, the pain control is not the best with these products. Oral transmucosal fentanyl citrate (OTFC) has been used successfully in treating breakthrough pain episodes associated with cancer. OTFC is a lozenge of fentanyl on a stick and is administered by continuously swabbing the interior of the subject's mouth until the product is dissolved (approximately 15 to 30 minutes). The buccal route of administration avoids the delay and variability associated with oral absorption.

BioDelivery Sciences International, Inc. (BDSI) has developed BEMA (BioErodible MucoAdhesive) fentanyl, an alternative product to OTFC that does not require the subject to continuously paint the inside of the mouth with the dosage form. The BDSI product is a small disc that is placed against the mucosal membrane inside the mouth. The mucoadhesive polymers in the disc readily adhere to the mucosal membrane (within 5 seconds) when moistened. The components of the disc are water soluble, so the entire dosage form dissolves within 30 minutes of application.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant and non-lactating female. A female of child-bearing potential is eligible to participate in this study if she is using an acceptable method of birth control.
* 18 years or older
* Patient must have pain associated with cancer or cancer treatment
* Patient must be on a stable current regimen of oral opioids equivalent to 60 - 1000 mg/day of oral morphine or 50 - 300 µg/hr of transdermal fentanyl (e.g. oxycodone 30 mg, methadone 20 mg, and hydromorphone 7.5 mg)
* Regularly experience 1 - 4 breakthrough pain episodes per day that require additional opioids for pain control
* At least partial relief of breakthrough pain by use of opioid therapy
* Subject must be able to self-administer the study medication correctly.
* Subject must be willing and able to complete the electronic diary card with each pain episode.
* Signed consent must be obtained at screening prior to any procedures being performed.

Exclusion Criteria:

* Psychiatric/cognitive or neurological impairment that would limit the subject's ability to understand or complete the diary
* Cardiopulmonary disease that, in the opinion of the investigator, would significantly increase the risk of respiratory depression
* Recent history or current evidence of alcohol or other drug substance (licit or illicit) abuse
* Rapidly escalating pain that the investigator believes may require an increase in the dosage of background pain medication during the study
* Moderate (Grade 3) to severe (Grade 4) mucositis (subjects with less than moderate mucositis are permitted and must be instructed to not apply the BEMA disc at a site of inflammation)
* Strontium 89 therapy within the previous 6 months
* Any other therapy prior to the study that the investigator considers could alter pain or the response to pain medication.
* Use of an investigational drug within 4 weeks preceding this study • History of hypersensitivity or intolerance to fentanyl
* Regularly more than 4 episodes per day
* ECOG performance status of 4 or 5
* Subject is pregnant, actively trying to become pregnant, breast feeding or not using adequate contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Blum, MD, Study Chair — BioDelivery Sciences International
Locations (1):
- ResearchPoint, Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment period was 3/14/06 - 6/13/08. Subjects were recruited from academic & private clinics in the US. Two groups of subjects were eligible for enrollment in this study. Subjects were eligible to enter this study following completion of the placebo-controlled study, FEN-201 or they were enrolled directly into this study.
Groups:
- Open Label Fentanyl Treatment: BioErodible Muco Adhesive(BEMA) Fentanyl
Period: Overall Study
Arm/Group | Open Label Fentanyl Treatment
Started | 244
Completed | 82
Not Completed | 162
Not completed — Withdrawal by Subject | 34
Not completed — Adverse Event | 30
Not completed — Death | 32
Not completed — Lack of Efficacy | 12
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 6
Not completed — Physician Decision | 21
Not completed — Other Reason | 22
Not completed — No dose taken | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label Fentanyl Treatment
Number analyzed (Participants) | 243
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 168
  >=65 years | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 58.0 (12.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 115
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 23
  White | 209
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  United States | 243

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events.
Description: After the first dose of BEMA Fentanyl, all adverse events were recorded and summarized.
Time Frame: Participants were followed for the duration of the study, an average of 126 days
Population: All subjects that received at least 1 dose of study drug were included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Open Label Fentanyl Treatment
Number analyzed (Participants) | 243
percentage of participants | 88.5

ADVERSE EVENTS:
Time Frame: The duration of a subject's particpation in the trial.
Description: From the start of study drug administration to the final follow-up visit.
Arm/Group | Open Label Fentanyl Treatment
Serious Adverse Events (participants affected / at risk) | 121/243
Other Adverse Events (participants affected / at risk) | 215/243
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Fentanyl Treatment (N=243)
anemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 3
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Haematemesis (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Chest pain (General disorders) | 1
Disease progression (General disorders) | 27
Implant site thrombosis (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pain (General disorders) | 2
Pyrexia (General disorders) | 2
Bile duct obstruction (Hepatobiliary disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Bronchitis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cellulitis orbital (Infections and infestations) | 1
Central line infection (Infections and infestations) | 1
Chest wall abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Intervertebral discitis (Infections and infestations) | 1
Klebsiella sepsis (Infections and infestations) | 1
Lung abscess (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 17
Pneumonia viral (Infections and infestations) | 1
Pseudomonal bacteraemia (Infections and infestations) | 1
Sepsis (Infections and infestations) | 5
Sepsis syndrome (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Accidental exposure (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Humerus fracture (Injury, poisoning and procedural complications) | 1
Cachexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Renal and urinary disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Adrenocortical carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Carcinoid syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cervix carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cervix neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hodgkin's disease recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian epithelial cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Recurrent cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Complicated migraine (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Mental status changes (Psychiatric disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 2
Urinary retention (Renal and urinary disorders) | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Reproductive system and breast disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Deep vein thrombosis (Vascular disorders) | 6
Haematoma (Vascular disorders) | 2
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open Label Fentanyl Treatment (N=243)
Anemia (Blood and lymphatic system disorders) | 31
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Abdominal Pain (Gastrointestinal disorders) | 14
Constipation (Gastrointestinal disorders) | 26
Diarrhoea (Gastrointestinal disorders) | 21
Dry mouth (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 74
Vomiting (Gastrointestinal disorders) | 52
Asthenia (General disorders) | 25
Disease progression (General disorders) | 28
Fatique (General disorders) | 25
Edema peripheral (General disorders) | 29
Pain (General disorders) | 22
Pyrexia (General disorders) | 25
Bronchitis (General disorders) | 13
Pheumonia (Infections and infestations) | 23
Urinary tract infection (Infections and infestations) | 16
Weight decreased (Investigations) | 15
Anorexia (Metabolism and nutrition disorders) | 16
Decreased appetite (Metabolism and nutrition disorders) | 18
Dehydration (Metabolism and nutrition disorders) | 29
Arthralgia (Musculoskeletal and connective tissue disorders) | 13
Back pain (Musculoskeletal and connective tissue disorders) | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16
Dizziness (Nervous system disorders) | 35
Headache (Nervous system disorders) | 24
Somnolence (Nervous system disorders) | 23
Anxiety (Psychiatric disorders) | 13
Confusional state (Psychiatric disorders) | 20
Depression (Psychiatric disorders) | 19
Insomnia (Psychiatric disorders) | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 16
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less